CLINICAL TRIAL: NCT02015468
Title: The Value of Early Mobilization and Physiotherapy Following Wrist Fractures Treated by Volar Plating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Ola-Lars Hammer, PhD-student, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1393A
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Distal Radius Fracture; Wrist Fracture
Keywords: Distal radius fracture; Wrist fracture; Physiotherapy; Immobilization; Volar locking plates; Mobilization
MeSH Terms: conditions — Wrist Fractures | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobilization (Experimental)
  Interventions: Other: Early mobilization
- Late mobilization (Experimental)
  Interventions: Other: Late mobilization

INTERVENTIONS:
Other: Early mobilization — Early weightbearing and physiotherapy
  Arms: Early mobilization
Other: Late mobilization — Late mobilization, none-weightbearing and home exercises
  Arms: Late mobilization

SUMMARY:
A prospective, randomized study investigating the possible benefits of immediate mobilization and frequent physiotherapy following a wrist fracture treated by volar plating.

The current study will test the following null hypothesis:

There is no significant difference between patients who receive a cast for the first 2 weeks postoperatively and then instructions in home exercises and patients who receive a cast for 2-3 days postoperatively and then have frequent sessions with a physiotherapist following volar locked plating for a extraarticular distal radius fracture, as evaluated by self-reported satisfaction after 3 months.

DETAILED DESCRIPTION:
The study will focus on patients treated with volar locked plating following an extraarticular distal radius fracture.

In a prospective manner the investigators intend to analyze hand function, x-ray and other parameters in order to investigate whether early mobilization and a targeted program of physiotherapy postoperatively leads to a better functional result and earlier return to a normal activity level. The investigators analysis will also focus on the safety of early mobilization with regards to possible detrimental effects on the osteosynthesis, bony union, associated soft-tissue injuries and functional outcome. The investigators also intend to assess the cost of more intensive follow-up and physiotherapy and do a cost-benefit evaluation.

ELIGIBILITY:
Inclusion Criteria:

Position prior to primary reduction:

* Dorsal tilt > 25°
* Radial shortening> 6 mm
* Radial inclination reduced by more than 15°
* Radiocarpal malalignment > 7 mm
* Dorsal /volar metaphyseal comminution
* Volar displacement of the distal fragment(= Smith's fracture)

Position after initial reduction:

* Dorsal tilt > 5°
* Radial shortening > 4 mm
* Radial inclination reduced by more than 10°
* Radiocarpal malalignment > 4 mm

Exclusion Criteria:

1. Gustilo-Anderson type III open fractures
2. Previous distal radius/ulna-fracture and/or disabling hand injury of the same extremity
3. Previous distal radius fracture or other disabling injury to the contralateral side
4. Dementia or other psychiatric illness which affect compliance
5. Congenital anomaly
6. Bilateral radius fracture
7. Concurrent fractures to the upper or lower extremities or other illness which affect movement of the extremities
8. Systemic joint disease such as rheumatoid arthritis
9. Patients who do not speak Norwegian
10. Pathological fracture other than osteoporotic fracture
11. Congenital bone disease (for example osteogenesis imperfecta)
12. Age below 18 and above 70
13. Patients not belonging to Akershus University Hospital

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-01-15 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Short version of "Disabilities of the Arm, Shoulder and Hand" (Quick-DASH) | 2 years
  The Quick-DASH score is a measure of patient reported satisfaction score and is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone.
Short Form 36 (SF36) | 2 years
  The SF-36 score is a quality of life measure and is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 2 years
  The PRWE-score is a measure of patient reported satisfaction and is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone
Euro-Qol 5 dimension score (EQ-5d) | 2 years
  The EQ-5d score is a quality of life measure and is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone
Pain Scores on the Visual Analog Scale (VAS) | 2 years
  The VAS-score is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone
Radiological findings (X-ray) | 2 years
  Angles, incongruity and other radiological parameters are compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone
Range of motion (ROM) | 2 yars
  Wrist range of motion is compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone
Cost analysis | 2 years
  The cost of treatment, sick-leave, complications and other socioeconomical parameters are compared between the group receiving early mobilization, weightbearing and physical therapy and the group receiving late mobilization and home exercises alone

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Madsen, Professor, Study Director — Oslo University Hospital
Locations (1):
- Akershus University Hospital, Oslo, Lorenskog, Norway